CLINICAL TRIAL: NCT05312450
Title: Integrated Traditional Chinese Medicine and Nutrition Treatments for Diabetes Care Cohort
Brief Title: TCM and Nutrition for Diabetes Care Cohort
Acronym: TCM-Nut-DC
Status: Completed | Type: Observational
Sponsor: Westlake University (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20211117ZJS001
Record Dates: First submitted 2021-12-02; First posted 2022-04-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Diabetes
Keywords: Diabetes; Nutrition; Gut microbiome; Metabolomics; Traditional Chinese medicine
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen including fecal, saliva, fasting boold, and fasting urine samples will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective cohort study that takes place in a clinic of Hangzhou, China. The aim of this study is to explore the molecular mechanism of special Chinese medicine formula combined with personalized nutrition to assist the treatment of diabetes from the aspect of multi-omics view. This study also aims to explore the relationship between gut microbiome and blood glucose in the process of personalized diet intervention.

DETAILED DESCRIPTION:
Traditional Chinese medicine has a history of more than two thousand years in China for treating diabetes based on the theory of "medicine and food homology". Modern pharmacological research and clinical research have shown that proprietary Chinese medicines and Chinese herbal decoctions have the advantages of overall regulation and fewer side effects for the treatment of type 2 diabetes and its complications. Meanwhile, dietary intervention is essential for the treatment of diabetes. In a clinic of Hangzhou, China, Chinese medicine doctors use a special Chinese medicine formula combined with dietary intervention to treat diabetes, and achieve good therapeutic effects without obvious adverse effects. The diet treatment plan is based on the results of the patient's food tolerance test, and dietary recommendations are provided based on the food glycemic index. In the first week of the treatment, patients are limit carbohydrate intake. Patients are evaluated every one month, and are instructed to choose foods rich in fiber and low glycemic index to reduce blood sugar fluctuations. Every patient is followed by one nutritionist, who provides dietary instructions for the patient. Patients use fingertip blood glucose to detect postprandial blood glucose. One course of treatment is three months, all patients will be treated for one course in this study. During the treatment, the dosage of western medicine hypoglycemic drugs was adjusted according to the Chinese Diabetes Prevention and Control Guidelines. Both Chinese medicine prescriptions and nutrition prescriptions were followed for the treatment to work towards the direction of drug injections-only oral drugs-drug reduction-drug discontinuation-drug discontinuation and stability-cure. Baseline information of demography, lifestyle, diet, physical activity, comorbidity, medication history, and so on is collected when patients enter the clinic to receive treatments. Meanwhile, the saliva, stool, fasting blood, fasting urine samples are collected. During the treatment, the dietary information is collected through photos taken by patients themselves. The saliva, stool, fasting blood, fasting urine samples are also collected when the patients re-enter the clinic for reexamination at the first week, and every one month.

ELIGIBILITY:
Inclusion Criteria:

* Comply with the diagnosis of diabetes in western medicine and the diagnostic criteria of type 2 diabetes in the "Guiding Principles for Clinical Research of New Chinese Medicines"; volunteer to participate and sign the informed consent form.

Exclusion Criteria:

* Major special diseases, such as mental system diseases or other cognitive impairment, cancer and other malignant wasting diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes who are volunteer to participate and sign the informed consent form, and without special diseases, such as mental system diseases or other cognitive impairment, cancer and other malignant wasting diseases.
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
gut microbiome | Baseline
  Fecal microbiome will be analyzed by metagenome sequencing
gut microbiome | The first week
  Fecal microbiome will be analyzed by metagenome sequencing
gut microbiome | The first month
  Fecal microbiome will be analyzed by metagenome sequencing
gut microbiome | The second month
  Fecal microbiome will be analyzed by metagenome sequencing
gut microbiome | The third month
  Fecal microbiome will be analyzed by metagenome sequencing
The change of postprandial blood glucose | Up to three months
  Fingertip blood glucose was used to detect postprandial blood glucose. The change of postprandial blood glucose among the three months will be measured

SECONDARY OUTCOMES:
Fecal metabolomics | Baseline
  Targeted or untargeted fecal metabolomics are performed
Fecal metabolomics | The first week
  Targeted or untargeted fecal metabolomics are performed
Fecal metabolomics | The first month
  Targeted or untargeted fecal metabolomics are performed
Fecal metabolomics | The second month
  Targeted or untargeted fecal metabolomics are performed
Fecal metabolomics | The third month
  Targeted or untargeted fecal metabolomics are performed
Serum metabolomics | Baseline
  Targeted or untargeted serum metabolomics are performed
Serum metabolomics | The first week
  Targeted or untargeted serum metabolomics are performed
Serum metabolomics | The first month
  Targeted or untargeted serum metabolomics are performed
Serum metabolomics | The second month
  Targeted or untargeted serum metabolomics are performed
Serum metabolomics | The third month
  Targeted or untargeted serum metabolomics are performed

CONTACTS AND LOCATIONS:
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China